CLINICAL TRIAL: NCT03017677
Title: The Establishment of a Cross-specialty Collaboration Platform Among Different Medical Specialties Based on High-risk Criteria for Mucopolysaccharidosis Confirmative Diagnosis
Brief Title: A Cross-specialty Collaboration Platform for Mucopolysaccharidosis Confirmative Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 16MMHIS127
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Mucopolysaccharidoses
MeSH Terms: conditions — Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group

SUMMARY:
In this study the investigators is aimed to establish the MPS screening algorithm for high risk patients who had medical history of previous surgical repair or presence of inguinal and/or umbilical hernia with combination of any ENT related surgery or examination in Taiwan.

DETAILED DESCRIPTION:
Mucopolysaccharidoses (MPS) are a group of inherited lysosomal storage disorders. In individuals with MPS disorders, have deficiency or malfunction of specific lysosomal enzymes leads to an abnormal accumulation of certain complex carbohydrates (mucopolysaccharides or glycosaminoglycans) in the arteries, skeleton, eyes, joints, ears, skin, and/or teeth. These accumulations may also be found in the respiratory system, liver, spleen, central nervous system, blood, and bone marrow. This accumulation eventually causes progressive damage to cells, tissues, and various organ systems of the body. Due to such an extreme variability in clinical presentation as well as wide range of disease spectrum, but insufficient MPS disease awareness in Taiwan, these resulted in a delay diagnosis or even miss diagnosis with other clinical symptom thus patient often received inappropriate treatment. In order to address the current issue of delay diagnosis among MPS patient, it is critical to develop a MPS screening algorithm for high risk patients in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 0-20 years of age.
* The subject had medical history of previous surgical hernia repair or presence of inguinal and/or umbilical hernia.
* The subject had or is scheduled for ENT surgery for any of the following, alone or in combination with adenoidectomy, tonsillectomy, ear tube insertion/tympanostomy, tracheotomy and bronchoscopy
* The subject who is willing and able to provide written, signed informed consent, or by a legally authorized representative after the nature of the study has been explained and prior to any research-related procedures.

Exclusion Criteria:

-The subject has a current confirmed diagnosis of any MPS disorder.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High risk MPS patient
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the positive screening rate of MPS subject (I, II VI and IV) under ENT screening algorithm in Taiwan | 3 Years

SECONDARY OUTCOMES:
To evaluate the data collection of patient profile which include urine GAG data, disaccharides patterns, enzyme activity, genetic pattern and medical history of MPS (I, II VI and IV) patients. | 3 Years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arn P, Bruce IA, Wraith JE, Travers H, Fallet S. Airway-related symptoms and surgeries in patients with mucopolysaccharidosis I. Ann Otol Rhinol Laryngol. 2015 Mar;124(3):198-205. doi: 10.1177/0003489414550154. Epub 2014 Sep 11. PMID 25214650
- [Result] Chuang CK, Lin HY, Wang TJ, Tsai CC, Liu HL, Lin SP. A modified liquid chromatography/tandem mass spectrometry method for predominant disaccharide units of urinary glycosaminoglycans in patients with mucopolysaccharidoses. Orphanet J Rare Dis. 2014 Sep 2;9:135. doi: 10.1186/s13023-014-0135-3. PMID 25178307
- [Result] Chuang CK, Lin SP, Chung SF. Diagnostic screening for mucopolysaccharidoses by the dimethylmethylene blue method and two dimensional electrophoresis. Zhonghua Yi Xue Za Zhi (Taipei). 2001 Jan;64(1):15-22. PMID 11310367
- [Result] Lin HY, Chen MR, Chuang CK, Chen CP, Lin DS, Chien YH, Ke YY, Tsai FJ, Pan HP, Lin SJ, Hwu WL, Niu DM, Lee NC, Lin SP. Enzyme replacement therapy for mucopolysaccharidosis VI--experience in Taiwan. J Inherit Metab Dis. 2010 Dec;33 Suppl 3:S421-7. doi: 10.1007/s10545-010-9212-5. Epub 2010 Oct 6. PMID 20924685
- [Result] Lin HY, Chuang CK, Wang CH, Chien YH, Wang YM, Tsai FJ, Chou YY, Lin SJ, Pan HP, Niu DM, Hwu WL, Ke YY, Lin SP. Long-term galsulfase enzyme replacement therapy in Taiwanese mucopolysaccharidosis VI patients: A case series. Mol Genet Metab Rep. 2016 Apr 18;7:63-9. doi: 10.1016/j.ymgmr.2016.04.003. eCollection 2016 Jun. PMID 27134829
- [Result] Neufeld EF, Muenzer J. The mucopolysaccharidoses. In: Scriver CR, Beaudet AL, Sly WS, Valle D, editors; Childs B, KinzlerKW, Vogelstein B, assoc. editors. The metabolic and molecular bases of inherited disease, 8th edition. New York: McGraw-Hill; 2001. pp 3421-52.
- [Result] Chuang CK, Lin SP. Neurochemical changes and therapeutical approaches in mucopolysaccharidoses. In: Sankar S, Michael A, Maheep B, editors. Neurochemistry of metabolic diseaseslysosomal storage diseases, phenylketouria and Canavan disease. Trivandrum, Kerala, India: Transworld Research Network; 2007. pp 1-20.